CLINICAL TRIAL: NCT02647047
Title: Spinal Analgesia Versus Epidural Analgesia in Minor Laparotomic Liver Surgery in an Enhanced Recovery Programme: A Randomized Controlled Trial
Brief Title: Spinal Versus Epidural Analgesia in Laparotomic Liver Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Elena Bignami, M.D., Ospedale San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VAS-LIVER
Record Dates: First submitted 2015-12-15; First posted 2016-01-06 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2016-01

CONDITIONS: Secondary Malignant Neoplasm of Liver; Liver Diseases; Liver Neoplasms
Keywords: spinal analgesia; epidural analgesia; laparotomic liver resection; ERAS; length of stay
MeSH Terms: conditions — Liver Diseases; Liver Neoplasms | interventions — Analgesia, Epidural; Acetaminophen; Ketorolac; Ropivacaine; Sufentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Spinal (Experimental): Patients will receive spinal analgesia (morphine 0.2 mg) before general anesthesia for minor laparotomic liver resection.
  Interventions: Procedure: Spinal analgesia; Procedure: Transversus Abdominis Plane block; Procedure: Surgical wound infiltration; Drug: Acetaminophen; Drug: Ketorolac; Drug: Ropivacaine
- Epidural (Active Comparator): Patients will receive epidural analgesia (bolus of ropivacaine 0.2% 4-6 mL followed by continuous epidural infusion of ropivacaine 0.2% 99 mL + sufentanil 50 mcg/mL 1 mL) before general anesthesia for minor laparotomic liver resection.
  Interventions: Procedure: Epidural analgesia; Drug: Acetaminophen; Drug: Ketorolac; Drug: Ropivacaine; Drug: Sufentanil

INTERVENTIONS:
Procedure: Spinal analgesia — Administration of morphine 0.2 mg in subarachnoid space.
  Arms: Spinal
Procedure: Epidural analgesia — Bolus of ropivacaine 0.2% 4-6 mL followed by continuous epidural infusion of ropivacaine 0.2% 99 mL + sufentanil 50 mcg/mL 1 mL in epidural space
  Arms: Epidural
Procedure: Transversus Abdominis Plane block — Administration of ropivacaine 0.375% 20 mL in the plane between the internal oblique and the transversus abdominis muscles, bilaterally
  Arms: Spinal
Procedure: Surgical wound infiltration — Infiltration of the surgical wound with ropivacaine 0.75% 10- 20 mL
  Arms: Spinal
Drug: Acetaminophen — Administration of 1000 mg of acetaminophen 40 minutes before ending of surgery followed by intravenous administration of 1000 mg every 8 hours
Drug: Ketorolac — Administration of a non-steroidal antinflammatory drug (ketorolac 30 mg) as a rescue therapy
Drug: Ropivacaine — Epidural bolus of ropivacaine 0.2% 4-6 mL followed by continuous epidural infusion of ropivacaine 0.2% 99 mL
  Arms: Epidural
Drug: Sufentanil — Epidural continuous epidural infusion of sufentanil 50 mcg/mL 1 mL
  Arms: Epidural
Drug: Ropivacaine — Administration of ropivacaine 0.375% 20 mL in the plane between the internal oblique and the transversus abdominis muscles, bilaterally to obtain the transversus abdominis plane block
  Arms: Spinal
Drug: Ropivacaine — Infiltration of the surgical wound with ropivacaine 0.75% 10- 20 mL
  Arms: Spinal

SUMMARY:
The purpose of this study is to evaluate the efficacy of spinal analgesia for minor laparotomic hepatectomy compared with epidural analgesia, monitoring visual analog scale (VAS). The investigators expect at least the same post-operative pain control in the two groups (non inferiority of pain control with spinal analgesia compared to epidural analgesia). Second endpoint is to verify whether after spinal analgesia there is a decrease in patient's length of hospitalization according to enhanced recovery after surgery (ERAS) principles.

DETAILED DESCRIPTION:
Liver surgery is performed under general anesthesia. Loco-regional analgesia is generally performed before general anesthesia induction to obtain the best post-operative pain control,in association with intravenous analgesic drug administration.

For minor laparotomic surgery (defined as the resection of up to three hepatic segments), if not contraindicated, in our hospital loco-regional analgesia is performed through the placement of a thoracic (T7-T8 or T8-T9) epidural catheter in which a local anesthetic (usually ropivacaine) and an opioid (usually sufentanil) are administered for the first three post-operative days. This is still considered the gold-standard for pain management in this surgery. In our institute, there is a dedicated acute pain service (APS) for pain management in the post-operative period. APS is also responsible for monitoring, registering and treating all side effects related to both the procedure and the drugs used.

In laparoscopic abdominal surgery, instead of epidural analgesia, if not contraindicated, spinal analgesia with low dose morphine before general anesthesia induction is performed. This technique is actually considered efficacy and safe in these type of surgeries.

The investigators therefore decided to test the efficacy of spinal analgesia versus epidural analgesia for minor liver surgery since anterior hepatic segments resection is less painful than major liver surgery because it requires less liver manipulation without significant involvement of the Glisson's capsule. This might imply a less incidence of procedure-related side effects such as post-dural puncture headache or site infections. Moreover, spinal analgesia may allow a earlier post-operative patients mobilization and thus a earlier hospital discharge.

In this randomized controlled trial, the investigators therefore aim to randomize 40 consecutive patients into 2 arms. The experimental group will receive spinal analgesia (morphine 0.2 mg) for post-operative pain control while the control group will receive epidural analgesia (bolus of ropivacaine 0.2% 4-6 mL followed by continuous epidural infusion of ropivacaine 0.2%: 99 mL + sufentanil 50 mcg/mL: 1 mL).

Randomization will be performed with closed opaque envelopes. During surgery, patients will be monitored as usual. Intraoperative blood losses and fluids administration will be recorded.

Patients randomized into the epidural group will not receive local anesthetic administration through the epidural catheter during the hepatic resection phase to avoid hemodynamic instability. Once the hepatic resection phase is finished and euvolemic status is recovered, epidural analgesia will be administered as mentioned before.

In patients in the spinal group, transversus abdominis plane (TAP) block with ropivacaine 0.375% 20 mL bilaterally or surgical wound infiltration with ropivacaine 0.75% 10- 20 mL will also be performed before anesthesia recovery.

In both groups, post-operative pain control will be managed with intravenous acetaminophen 1000 mg 40 minutes before ending of surgery followed by intravenous administration of acetaminophen 1000 mg every 8 hours and a non-steroidal antinflammatory drug (ketorolac 30 mg) as a rescue therapy in the post-operative period if not contraindicated.

Patients will be monitored every 24 hours until the achievement of the "ready to discharge" status defined as:

* appropriate oral alimentation;
* optimal pain control with drugs administered orally;
* adequate ability in walking and personal care;
* clinical, laboratory and instrumental absence of any post-operative complication;
* intestinal function recovery;
* patient consent to discharge.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Hospitalized patients
* Surgical indication for minor laparotomic anterior liver resection (II, III, IV and V hepatic segment resection)
* Surgical indication for laparotomic liver metastasectomy
* Ability to provide an informed consent

Exclusion Criteria:

* Patient refusal to provide informed consent
* Chronical therapy with opioids
* Pregnancy or breastfeeding
* Alcohol or drug abuse
* Planned or unplanned post-operative intensive care unit admission
* Contraindication to spinal/epidural analgesia
* Severe liver or renal failure
* Cognitive disorders, mental retard or psychiatric disorders
* Allergy to any drug used

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of postoperative pain control by mean of the visual analog scale early after surgery | Within 1 hour after surgery
  Visual analog scale (VAS) will be assessed and compared between the two groups.
Assessment of postoperative pain control by mean of the visual analog scale six hours after surgery | 6 hours after surgery
  Visual analog scale (VAS) will be assessed and compared between the two groups.
Assessment of postoperative pain control by mean of the visual analog scale one day after surgery | 24 hours after surgery
  Visual analog scale (VAS) will be assessed and compared between the two groups.
Assessment of postoperative pain control by mean of the visual analog scale two days after surgery | 48 hours after surgery
  Visual analog scale (VAS) will be assessed and compared between the two groups.
Assessment of postoperative pain control by mean of the visual analog scale three days after surgery | 72 hours after surgery
  Visual analog scale (VAS) will be assessed and compared between the two groups.
Assessment of postoperative pain control by mean of the visual analog scale at hospital discharge | Up to 30 days after surgery
  Visual analog scale (VAS) will be assessed and compared between the two groups.

SECONDARY OUTCOMES:
Ready to discharge status | Up to 30 days after surgery
  The postoperative day in which patients reach the "ready to discharge" status will be recorded and compared between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Raffaella Reineke, M.D., Principal Investigator — Ospedale San Raffaele
Locations (1):
- Ospedale San Raffaele, Milan, MI, Italy

REFERENCES:
- [Background] Tzimas P, Prout J, Papadopoulos G, Mallett SV. Epidural anaesthesia and analgesia for liver resection. Anaesthesia. 2013 Jun;68(6):628-35. doi: 10.1111/anae.12191. PMID 23662750
- [Background] Revie EJ, Massie LJ, McNally SJ, McKeown DW, Garden OJ, Wigmore SJ. Effectiveness of epidural analgesia following open liver resection. HPB (Oxford). 2011 Mar;13(3):206-11. doi: 10.1111/j.1477-2574.2010.00274.x. PMID 21309939
- [Background] Kasivisvanathan R, Abbassi-Ghadi N, Prout J, Clevenger B, Fusai GK, Mallett SV. A prospective cohort study of intrathecal versus epidural analgesia for patients undergoing hepatic resection. HPB (Oxford). 2014 Aug;16(8):768-75. doi: 10.1111/hpb.12222. Epub 2014 Jan 28. PMID 24467320
- [Background] Ntinas A, Kardassis D, Konstantinopoulos I, Kottos P, Manias A, Kyritsi M, Zilianiaki D, Vrochides D. Duration of the thoracic epidural catheter in a fast-track recovery protocol may decrease the length of stay after a major hepatectomy: a case control study. Int J Surg. 2013;11(9):882-5. doi: 10.1016/j.ijsu.2013.07.014. Epub 2013 Aug 4. PMID 23924906
- [Background] Koea JB, Young Y, Gunn K. Fast track liver resection: the effect of a comprehensive care package and analgesia with single dose intrathecal morphine with gabapentin or continuous epidural analgesia. HPB Surg. 2009;2009:271986. doi: 10.1155/2009/271986. Epub 2009 Dec 15. PMID 20029637
- [Background] Hughes MJ, McNally S, Wigmore SJ. Enhanced recovery following liver surgery: a systematic review and meta-analysis. HPB (Oxford). 2014 Aug;16(8):699-706. doi: 10.1111/hpb.12245. Epub 2014 Mar 24. PMID 24661306